CLINICAL TRIAL: NCT03249246
Title: Epidemiology of Sepsis in Turkish ICUs :a National Point Prevalence Multi-centre Study.
Brief Title: Epidemiology of Sepsis in Turkish ICUs.
Status: Completed | Type: Observational
Sponsor: Nur Baykara (Other)
Collaborators: Turkish Society of Intensive Care, Sepsis Study Group (Unknown)
Responsible Party: Sponsor-Investigator, Nur Baykara, Prof.Dr.Nur Baykara, Turkish Intensive Care Society
Organization: Turkish Intensive Care Society (Other)
Other Study IDs: TurkishICS
Record Dates: First submitted 2017-08-09; First posted 2017-08-15 (Actual); Last update posted 2017-08-15 (Actual); Status verified 2017-08

CONDITIONS: Sepsis; Septic Shock; Severe Sepsis
Keywords: Sepsis; ICU; Point prevalence
MeSH Terms: conditions — Sepsis; Shock, Septic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Infection only: The patients have only infection
  Interventions: Other: No intervention
- Infection + SIRS: Patients have infection plus systemic inflammatory response syndrome (SIRS)
  Interventions: Other: No intervention
- Severe sepsis: Septic patients with newly developed organ dysfunctions
  Interventions: Other: No intervention
- Septic shock: Sepsis plus sepsis related hypotension
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention

SUMMARY:
The prevalence and mortality of sepsis in Turkey is not know at large. Turkish Society of Intensive Care Medicine, Sepsis Study Group conducted a multi-centre,point prevalence survey to determine the prevalence, causative micro-organisms and outcome of sepsis in Turkish ICUs.

ELIGIBILITY:
Inclusion Criteria:All patients present on or admitted to participating ICU on study day.

Exclusion Criteria:

* Age<18 years
* Patients who underwent cardiovascular surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients (>18 yr)present on the participating ICU or admitted to participating ICUs on study day
Sampling Method: Probability Sample
Enrollment: 1499 (Actual)
Dates: Start 2016-01-27 (Actual); Primary Completion 2016-01-28 (Actual); Study Completion 2016-02-27 (Actual)

PRIMARY OUTCOMES:
Prevalence of sepsis | Up to 12 weeks.
  The prevalence of sepsis,Severe sepsis and septic shock on study day

SECONDARY OUTCOMES:
Mortality rate of sepsis | Mortality at 30 days
  Mortality rate of septic shock

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rhodes A, Phillips G, Beale R, Cecconi M, Chiche JD, De Backer D, Divatia J, Du B, Evans L, Ferrer R, Girardis M, Koulenti D, Machado F, Simpson SQ, Tan CC, Wittebole X, Levy M. The Surviving Sepsis Campaign bundles and outcome: results from the International Multicentre Prevalence Study on Sepsis (the IMPreSS study). Intensive Care Med. 2015 Sep;41(9):1620-8. doi: 10.1007/s00134-015-3906-y. Epub 2015 Jun 25. PMID 26109396
- [Background] Falagas ME, Rafailidis PI, Kofteridis D, Virtzili S, Chelvatzoglou FC, Papaioannou V, Maraki S, Samonis G, Michalopoulos A. Risk factors of carbapenem-resistant Klebsiella pneumoniae infections: a matched case control study. J Antimicrob Chemother. 2007 Nov;60(5):1124-30. doi: 10.1093/jac/dkm356. Epub 2007 Sep 20. PMID 17884829
- [Result] Fleischmann C, Scherag A, Adhikari NK, Hartog CS, Tsaganos T, Schlattmann P, Angus DC, Reinhart K; International Forum of Acute Care Trialists. Assessment of Global Incidence and Mortality of Hospital-treated Sepsis. Current Estimates and Limitations. Am J Respir Crit Care Med. 2016 Feb 1;193(3):259-72. doi: 10.1164/rccm.201504-0781OC. PMID 26414292
- [Derived] Baykara N, Akalin H, Arslantas MK, Hanci V, Caglayan C, Kahveci F, Demirag K, Baydemir C, Unal N; Sepsis Study Group. Epidemiology of sepsis in intensive care units in Turkey: a multicenter, point-prevalence study. Crit Care. 2018 Apr 16;22(1):93. doi: 10.1186/s13054-018-2013-1. PMID 29656714